CLINICAL TRIAL: NCT05747365
Title: Cross-sectional Case-control Study on the Role of Endocrine Disruptors in Thyroid Cancer
Brief Title: Role of Endocrine Disruptors in Thyroid Cancer
Acronym: THY-ED
Status: Recruiting | Type: Observational
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Other Study IDs: 05C214
Record Dates: First submitted 2023-02-17; First posted 2023-02-28 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Endocrine Disruptor Chemicals; Thyroid Cancer
MeSH Terms: conditions — Thyroid Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case group: Patients with thyroid cancer diagnosis within 5 years before study enrollment
  Interventions: Diagnostic Test: Blood and urine diagnostic evaluation
- Control group: Patients without clinical diagnosis of thyroid disease
  Interventions: Diagnostic Test: Blood and urine diagnostic evaluation

INTERVENTIONS:
Diagnostic Test: Blood and urine diagnostic evaluation — Blood and urine samples will be obtained from both case and control groups in order to evaluate EDCs concentrations

SUMMARY:
the relationship between human exposure to EDCS and TC is poorly investigated and still unclear. The aim of this study is to evaluate the possible role of old and new generation endocrine disruptors in thyroid cancer. The primary aim is to evaluate the difference in the average levels of the main endocrine disruptors (PFAS, including: PFOA, PFOS, PFDA, PFUnA, PFHpS and possibly subsequently other categories, such as bisphenols, phthalates, parabens, PCBs, flame retardants) between patients with and without a diagnosis of thyroid cancer through highly sensitive, selective and precise mass spectrometry methods, such as liquid chromatography combined with tandem mass spectrometry (LC-MS / MS).

The secondary aim is to evaluate the relationship between the concentrations of endocrine disruptors and some anamnestic variables studied (for example the type of diet, the use of personal care products).

ELIGIBILITY:
Inclusion Criteria:

* patients with a diagnosis of thyroid cancer in the last 5 years (arm A)
* patients without a diagnosis of thyroid cancer will match patients included in arm A

Exclusion Criteria:

* subjects under 18 years old
* patients unable to sign the informed consent or questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all patients referred to our tertiary clinical center for thyroid cancer diagnosed in the last 5 years will be consecutively enrolled (case population). Patients without a diagnosis of thyroid cancer will match patients included in the case population, according to age and sex.
Sampling Method: Non-Probability Sample
Enrollment: 222 (Estimated)
Dates: Start 2022-07-12 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Difference in the average levels of the main endocrine disruptors | At recruitment
  The main endocrine disruptors evaluated will be PFAS, including: PFOA, PFOS, PFDA, PFUnA, PFHpS and possibly subsequently other categories, such as bisphenols, phthalates, parabens, PCBs, flame retardants
Relationship between the concentrations of endocrine disruptors and anamnestic variables | At recruitment
  Relationship between the concentrations of endocrine disruptors and some anamnestic variables studied (for example the type of diet, the use of personal care products).

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Auxologico Italiano, IRCCS, Milan, Italy